CLINICAL TRIAL: NCT00876096
Title: Development and Validation of Fungal Extraction and Real -Time PCR Assay for the Diagnosis of Medically Important Fungal Infections in Blood Samples.
Brief Title: Interest of Real-time Polymerase Chain Reaction (PCR) in the Diagnosis of Fungal Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-API-03
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2009-04

CONDITIONS: Healthy; Fungal Infections
Keywords: Diagnosis, Differential
MeSH Terms: conditions — Mycoses; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): precocious diagnosis and taken care therapeutics of the systematic athlete's feet
  Interventions: Other: Catch of blood then PCR

INTERVENTIONS:
Other: Catch of blood then PCR — To optimize the technology of extraction of nucleic acids of origin fongique by collaborating with the laboratories of Parasitologie and Mycology of the TEACHING HOSPITAL of Rennes and Toulouse.

SUMMARY:
Invasive fungal infections have a major impact on the morbidity and mortality of immunocompromised patients, including patients with hematological malignancies, neutropenic patients, human immunodeficiency virus infected patients, diabetics, solid organ transplanted patients and patients admitted in an intensive care unit.

The survival of these patients depends on early diagnosis and prompt appropriate antifungal treatment. The early diagnosis of these infections is difficult because of the lack of sensitive test methods, notably blood cultures. For these reasons, the investigators decided to develop a real-time PCR (Polymerase Chain Reaction) assay on blood samples. It should allow rapid response to establish a positive or negative diagnosis of invasive fungal infection, could contribute strongly to the decision of treating using antifungals, and should monitor the effectiveness and the optimization of antifungal prescriptions.

The investigators' objectives are: First, to validate an extraction method from blood infected by fungi species. Secondly, the investigators want to develop three real-time PCR: A fungal real-time PCR able to detect most fungal species; a real-time PCR targetting Candida albicans and Aspergillus fumigatus which are two clinically important pathogens. Then blood samples of patients (classified according to EORTC consensus) will be collected during the study in order to evaluate and validate our method on clinical samples. Results will allow the investigators to determine the sensitivity, specificity and reproducibility, negative and predictive values.

Overall, the investigators' work aims to evaluate the clinical impact of real-time PCR in the early diagnosis of invasive fungal infections and on the initiation or stopping of antifungal therapy. The economic impact resulting from the use of this method will be evaluated.

DETAILED DESCRIPTION:
Invasive fungal infections are a major cause of morbidity and mortality in immunocompromised patients. Among them, patients with hematological malignancies, neutropenic patients, human immunodeficiency virus infected patients, diabetics, solid organ transplanted patients and patients admitted in an intensive care unit are particularly at high risk.

The survival of these patients depends on early diagnosis and prompt appropriate antifungal treatment. The early diagnosis of these infections is difficult because of the lack of sensitive test methods, notably blood cultures. Its sensitivity is poor or close-zero for aspergillosis. In addition, the response time is several days. For these reasons, we decided to develop a real-time PCR (Polymerase Chain Reaction) assay on blood samples. It should allow rapid response to establish a positive or negative diagnosis of invasive fungal infection, it could contribute strongly to the decision of treating using antifungals, and it should monitor the effectiveness and the optimization of antifungal prescriptions.

Methods:

Our project is a multicentre prospective inter-regional collaborative work between Nice, Rennes and Toulouse Mycological and parasitological laboratories. Our objectives are: First, to validate an extraction method from blood infected by fungi species. The three laboratories will work together to determine the best extraction method, since there is no consensus method for the extraction of nucleic acids of fungal origin in the context of human infections. The numerous extraction techniques already used lead to differences in the PCR results. As a consequence, inter-laboratory comparisons are not easy. Secondly, we aim to develop three real-time PCR assays: A panfungal real-time PCR assay able to detect most fungal species responsible for human diseases; a real-time PCR assay targetting Candida albicans and one targeting Aspergillus fumigatus which are two clinically important pathogens. Then patient blood samples (classified according to EORTC consensus) will be collected during the study in order to evaluate and validate our method on clinical samples. Results will allow us to determine the sensitivity, specificity and reproducibility, negative and predictive values.

Objectives Overall, our work aims to evaluate the clinical impact of real-time PCR in the early diagnosis of invasive fungal infections and on the initiation or stopping of antifungal therapy. The economic impact resulting from the use of this method will be evaluated. Indeed, an excellent predictive negative value of a panfungal real-time PCR assay could warrant a decrease in the use of empirical antifungal therapy

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: Chosen healthy subjects are donors of the Blood transfusion centre of NICE
* Ill subjects:

  * Medical examination compatible with inclusion to donate blood
  * To sign lit consent
  * Affiliation to the regime of French national health and pensions organization
  * Patient as whom there is intention to deal by systematic antifongique, Criteria, linked to the guest, clinical and microbiological are defined

Exclusion Criteria:

* Minor or person over 18 under tutelage.
* Subjects deprived of freedom.
* Patients cancelling their consent.
* Patients violating the research protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The evaluation will be conducted on blood samples inoculated with known concentrations of numerous fungal species (various Candida sp, various Aspergillus sp., Cryptococcus sp. etc…). Extraction method and PCR techniques | 1 year

SECONDARY OUTCOMES:
IN Nice, Rennes and Toulouse Teaching hospitals, patients suspected of invasive fungal infection will be included in order to classified in three categories: proven, probable and possible fungal infection, according to EORTC consensus. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MARTY Pierre, PhD, Principal Investigator — CHU de Nice - laboratoire de parasitologie- Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (4):
- France (4):
  - CAL, Nice, Alpes-maritimes
  - CHU de Nice - 4 avenue Reine Victoria, Nice, Alpes-Maritimes
  - CHU de Rennes, Rennes
  - CHU de Touloluse - hôpital de Rangueil, Toulouse